CLINICAL TRIAL: NCT06577103
Title: A Comparative Study Between the Analgesic Effect of Pericapsular Nerve Group Block (PENG) With Lateral Femoral Cutaneous Nerve Block (LFCN) and Pericapsular Nerve Group Block (PENG) With Supra-inguinal Fascia Iliaca Block (SIFIC) in Hip Hemiarthroplasty: a Prospective Randomized Clinical Trial
Brief Title: The Analgesic Effect of Pericapsular Nerve Group Block With Lateral Femoral Cutaneous Nerve Block and Pericapsular Nerve Group Block With Supra-inguinal Fascia Iliaca Block in Hip Hemiarthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Moussa Elsayed, Assistant Lecturer of Anesthesiology, Surgical Intensive Care and Pain Medicine, Ain Shams University,Egypt, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FMASU MD345/2023
Record Dates: First submitted 2024-08-27; First posted 2024-08-29 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-05

CONDITIONS: Pericapsular Nerve Group Block; Lateral Femoral Cutaneous Nerve Block; Supra-inguinal Fascia Iliaca Block; Hip Hemiarthroplasty

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pericapsular nerve group block (PENG) with supra-inguinal fascia iliaca block (SIFIC) (Experimental): Patients will receive pericapsular nerve group (PENG) block with supra-inguinal fascia iliaca (SIFIC) block.
  Interventions: Other: Pericapsular nerve group block (PENG) with supra-inguinal fascia iliaca block (SIFIC)
- Pericapsular nerve group block (PENG) with lateral femoral cutaneous nerve block (LFCN) (Experimental): Patients will receive pericapsular nerve group (PENG) block with lateral femoral cutaneous nerve (LFCN) block.
  Interventions: Other: Pericapsular nerve group block (PENG) with lateral femoral cutaneous nerve block (LFCN)

INTERVENTIONS:
Other: Pericapsular nerve group block (PENG) with supra-inguinal fascia iliaca block (SIFIC) — Patients will receive pericapsular nerve group (PENG) block with supra-inguinal fascia iliaca (SIFIC) block.
  Arms: Pericapsular nerve group block (PENG) with supra-inguinal fascia iliaca block (SIFIC)
Other: Pericapsular nerve group block (PENG) with lateral femoral cutaneous nerve block (LFCN) — Patients will receive pericapsular nerve group (PENG) block with lateral femoral cutaneous nerve (LFCN) block.
  Arms: Pericapsular nerve group block (PENG) with lateral femoral cutaneous nerve block (LFCN)

SUMMARY:
The aim of this study is to investigate the efficiency of preoperative and post-operative analgesia by pericapsular nerve group block (PENG) block with supra-inguinal fascia iliaca block (SIFIC) block compared with PENG block with lateral femoral cutaneous nerve block (LFCN) block in ease of giving a sitting position for spinal anesthesia and reducing narcotic consumption during the first 24 hour post-operatively and functional recovary by using the Visual analogue scale (VAS) of pain.

DETAILED DESCRIPTION:
The established practice to decrease pain using opioids in hip fracture surgery may result in compromised outcomes in the frail and elderly population with nausea-vomiting, constipation, delirium and respiratory depression. This popularized the regional analgesic techniques in the surgical treatment of hip fractures. Femoral nerve (FN) and supra-inguinal fascia iliaca block (SIFIC) block are documented to provide good peri-operative analgesia with reduced need for opioids.

The latest pericapsular nerve group block (PENG) block, is an interfacial plane block targeting the articular branches of the femoral, obturator (ON) and accessory obturator nerves (AON) at the hip.

An ability to perform in supine positioning, which is especially important in patients with acute hip fractures or chronic pain is an indigenous advantage of PENG block. Due to the blockade of only sensory articular branches, substantial motor weakness is unexpected. But exclusive use of PENG block for analgesia in hip fracture patients is not sufficient as it doesn't involve the cutaneous pain-generating area supplied by the lateral femoral cutaneous nerve block (LFCN).

ELIGIBILITY:
Inclusion Criteria:

* Age 40-80 years.
* Sex: Both sexes.
* American Society of Anaesthesiologists (ASA) Physical Status Class I, II, and III.
* Scheduled for hip hemiarthroplasty under general anesthesia.

Exclusion Criteria:

* Declining to give a written informed consent.
* History of allergy to the medications used in the study.
* Contraindications to regional anesthesia (including patient refusal, coagulopathy and local infection).
* Psychiatric disorders or narcotic abusers.
* Significant cognitive dysfunction.
* American Society of Anesthesiologists (ASA) Physical Status Class IV.
* Renal insufficiency (to avoid local anesthetic or nalbuphine metabolites adverse effect)
* Opioid abuser patients
* Pregnancy.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2024-01-02 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
Degree of pain | 24 hours postoperatively
  Degree of pain will be assessed by visual analogue score (VAS). VAS ranging from 0 to 10, where 0 is no pain and 10 is maximum pain. It will be assessed preoperatively first after the block application then postoperatively, at post anesthesia care unit (PACU) and then 2, 6 ,12 ,18 ,24 hours postoperatively.

SECONDARY OUTCOMES:
The ease of giving a sitting position for spinal anesthesia (EOSP) | Intraoperatively
  The ease of giving a sitting position for spinal anesthesia (EOSP) will be assessed by the EOSP score .EOSP was assessed on the scale of 0-3 (0 = unable to position, 1 = patient had abnormal posturing due to pain and required support for positioning, 2 = mild discomfort but does not require support for positioning, 3 = optimal condition where the patient was able to position himself
The total dose of nalbuphine consumption | 24 hours postoperatively
  When visual analogue score (VAS) >/=4, patients will receive injection nalbuphine 10 mg/70 kg (with maximum dose 160 mg over 24 hours) intravenously.
The number of patients who needed rescue analgesia | 24 hours postoperatively
  Number of patients who needed rescue analgesia will be recorded
Ablility to walk with support within 24 hours | 24 hours postoperatively
  The ability of patients to walk with support will be recorded

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.